CLINICAL TRIAL: NCT00460434
Title: Outcomes Following Vaginal Prolapse Repair and Mid Urethral Sling (OPUS) Trial
Brief Title: Outcomes Following Vaginal Prolapse Repair and Mid Urethral Sling Trial
Acronym: OPUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Collaborators: Office of Research on Women's Health (ORWH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15P01; 2U01HD041249 (NIH); 2U10HD041250 (NIH); 2U10HD041261 (NIH); 2U10HD041267 (NIH); 1U10HD054136 (NIH); 1U10HD054214 (NIH); 1U10HD054215 (NIH); 1U10HD054241 (NIH)
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: Prolapse; Urinary incontinence; TVT
MeSH Terms: conditions — Pelvic Organ Prolapse; Prolapse; Urinary Incontinence | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Tension-free Vaginal Tape (TVT) surgery
  Interventions: Device: TVT
- 2 (Sham Comparator): Sham Tension-free Vaginal Tape (TVT) surgery
  Interventions: Other: Sham

INTERVENTIONS:
Device: TVT — Prophylactic TVT
  Arms: 1
Other: Sham — Sham TVT
  Arms: 2

SUMMARY:
Pelvic organ prolapse is common among women with a prevalence that has been estimated to be as high as 30%. Prolapse may be corrected by surgery using either a vaginal or abdominal incision. Some women develop stress urinary incontinence (SUI) after surgery. A prior randomized trial has shown that use of a Burch sling at the time of an abdominal sacrocolpopexy decreases the risk of urinary incontinence; however, the benefit of adding an anti incontinence procedure to prevent SUI at the time of prolapse surgery performed via a vaginal approach is unclear. Thus, the objective of the Outcomes following vaginal Prolapse repair and mid Urethral Sling (OPUS) trial is to determine whether prophylactic treatment with Tension-free Vaginal Tape (TVT)® at the time of prolapse surgery done via a vaginal approach is effective in preventing urinary incontinence.

DETAILED DESCRIPTION:
The overall objective of this randomized clinical trial is to determine whether symptom-specific treatment of incontinence after prolapse surgery is equally effective to prophylactic treatment by adding TVT® at the time of the prolapse surgery among women with anterior vaginal prolapse but without pre-operative symptoms of stress urinary incontinence.

The primary aims are:

In stress continent women planning vaginal surgery for pelvic organ prolapse:

1. To determine if the failure rate defined by subsequent treatment for urinary incontinence, signs or symptoms of bothersome urinary incontinence [defined as having at least moderate bother for any of 4 Pelvic Floor Distress Inventory (PFDI) incontinence items] differs between vaginal prolapse repair and vaginal prolapse repair plus TVT® during the first 3 months after the index surgery.
2. To determine if the prevalence of bothersome urinary incontinence at 12 months after the index surgery differs between vaginal prolapse repair and vaginal prolapse repair plus TVT®, whether or not there was subsequent treatment for symptoms of urinary incontinence; i.e., to determine whether symptom-specific treatment of incontinence after prolapse surgery is equally effective to prophylactic treatment by adding a TVT® at the time of the prolapse surgery.
3. To measure the total cost of care and relate the difference in cost of care between the two groups to differences in health utilities and health-related quality of life, which will allow us to examine the cost-effectiveness of prophylactic use of a TVT® at the time of prolapse surgery versus symptom-specific treatment of stress incontinence after prolapse surgery.

ELIGIBILITY:
Inclusion Criteria:

Vaginal bulge symptoms as indicated by an affirmative response to either questions 4 or 5 of the PFDI:

* Do you usually have a sensation of bulging or protrusion from the vaginal area?
* Do you usually have a bulge or something falling out that you can see or feel in the vaginal area? Anterior vaginal prolapse defined by pelvic organ prolapse quantification (POP-Q) Point Aa ≥ -1 cm (i.e., -1,0,1,2, or 3 cm).

Surgical plan that includes a vaginal approach for apical or anterior prolapse repair.

Able and willing to complete data collection per protocol, including written informed consent.

Exclusion Criteria:

Pregnancy or planning pregnancy in the first postoperative year. Any prior mid urethral sling. Currently participating in another interventional study for urinary incontinence.

Untreated urinary tract infection (may be included after resolution).

Overt symptoms of stress urinary incontinence as defined by a positive response to any of the following 3 PFDI items:

* Do you usually experience urine leakage related to coughing, sneezing, or laughing?
* Do you usually experience urine leakage related to physical exercise such as walking, running, aerobics, or tennis?
* Do you usually experience urine leakage related to lifting or bending over? Currently being treated for stress urinary incontinence with pessary/incontinence ring, pelvic floor muscle exercise or medication (duloxetine and imipramine, and alpha agonists).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2007-05; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John T Wei, MD, Principal Investigator — University of Michigan
Locations (8):
- United States (8):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - USCD Medical Center, La Jolla, California
  - Kaiser Permanente, San Diego, California
  - Loyola University Medical Center, Maywood, Illinois
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - UT Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Wei JT, Nygaard I, Richter HE, Nager CW, Barber MD, Kenton K, Amundsen CL, Schaffer J, Meikle SF, Spino C; Pelvic Floor Disorders Network. A midurethral sling to reduce incontinence after vaginal prolapse repair. N Engl J Med. 2012 Jun 21;366(25):2358-67. doi: 10.1056/NEJMoa1111967. PMID 22716974
- [Derived] Baessler K, Christmann-Schmid C, Haya N, Mowat A, Chen Z, Wallace SA, Yeung E, Maher C. Surgery for women with pelvic organ prolapse with or without stress urinary incontinence. Cochrane Database Syst Rev. 2026 Feb 6;2(2):CD013108. doi: 10.1002/14651858.CD013108.pub2. PMID 41649019
- [Derived] Lukacz ES, Sridhar A, Chermansky CJ, Rahn DD, Harvie HS, Gantz MG, Varner RE, Korbly NB, Mazloomdoost D; Eunice Kennedy Shriver National Institute of Child Health and Human Development Pelvic Floor Disorders Network (PFDN). Sexual Activity and Dyspareunia 1 Year After Surgical Repair of Pelvic Organ Prolapse. Obstet Gynecol. 2020 Sep;136(3):492-500. doi: 10.1097/AOG.0000000000003992. PMID 32769645

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All women presenting to the participating PFDN clinical centers with the complaint of prolapse, as defined by the inclusion criteria, will be screened for the subjective complaint of SUI using items on the PFDI. Eligible individuals will be offered RCT participation.
Pre-assignment Details: Participants consisted of women who were being considered for an apical and/or anterior vaginal prolapse repair via a vaginal approach without subjective complaints of SUI. They must have had vaginal bulge symptoms (defined as positive responses to the PFDI), and anterior vaginal prolapse with point Aa at -1cm or greater (determined by POP-Q).
Groups:
- Midurethral Sling: Women in this arm received a concomitant tension-free vaginal tape (TVT) procedure.
- Sham Incision: Women in this arm received two one-centimeter suprapubic incisions, comparable to those received in the intervention group.
Period: Overall Study
Arm/Group | Midurethral Sling | Sham Incision
Started | 165 | 172
3 Months | 163 | 171
12 Months | 162 | 165
Completed | 162 | 165
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midurethral Sling | Sham Incision | Total
Number analyzed (Participants) | 165 | 172 | 337
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (10.8) | 62.2 (10.2) | 62.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 172 | 337
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 143 | 143 | 286
  Black | 10 | 14 | 24
  Asian | 3 | 2 | 5
  Other | 9 | 13 | 22
  Hispanic | 21 | 27 | 48
  Not Hispanic | 144 | 145 | 289
Annual Income <$30,000 [Count of Participants; unit: Participants] — Population: Self-reported question, population is those who provided a response.
  Participants
    number analyzed (Participants) | 64 | 65 | 129
    (all) | 31 | 27 | 58
Married [Count of Participants; unit: Participants] — Population: Self-reported question, population is those who provided a response.
  Participants
    number analyzed (Participants) | 163 | 161 | 324
    (all) | 121 | 101 | 222
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 27.8 (4.9) | 28.1 (5.5) | 28.0 (5.2)
Pelvic Organ Prolapse Quantification [Count of Participants; unit: Participants] — (1=lowest point of prolapse is >1cm above the hymen; 2=within 1 cm above or below the hymen; 3= >1cm below the hymen but protrudes no more than 2cm less than the total vaginal length; 4=complete vaginal eversion)
  Participants
    2 | 45 | 48 | 93
    3 | 107 | 106 | 213
    4 | 13 | 18 | 31
Positive Cough Stress Test [Count of Participants; unit: Participants] — A leakage of urine with coughing or straining in either the supine or standing position with the bladder filled through a urethral catheter to 300ml.
  Participants | 54 | 57 | 111
Anterior Vaginal - Prolapse Repair [Count of Participants; unit: Participants]
  Anterior Repair Only | 20 | 17 | 37
  Apical Suspension Only | 32 | 42 | 74
  Both Anterior Repair and Apical Suspension | 101 | 100 | 201
  Colpocleisis | 11 | 13 | 24
Posterior Vaginal - Prolapse Repair [Count of Participants; unit: Participants] | 74 | 80 | 154
Previous Hysterectomy [Count of Participants; unit: Participants] | 62 | 66 | 128
Concomitant Hysterectomy [Count of Participants; unit: Participants] | 82 | 83 | 165

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Failure Defined as Subsequent Treatment for Urinary Incontinence, Signs or Symptoms of Bothersome Urinary Incontinence
Description: Defined as a positive cough stress test, bothersome incontinence symptoms, or treatment for urinary incontinence, and urinary incontinence (stress, urge, or mixed), regardless of whether interim treatment for incontinence had been provided.
Time Frame: 3 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Midurethral Sling | Sham Incision
Number analyzed (Participants) | 165 | 172
Participants | 39 | 85

2. Primary Outcome: Prevalence of Bothersome Urinary Incontinence at 12 Months Following Index Surgery
Description: Defined as a positive cough stress test or report of bothersome incontinence symptoms.
Time Frame: 12 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Midurethral Sling | Sham Incision
Number analyzed (Participants) | 165 | 172
Participants | 45 | 74

3. Secondary Outcome: Medical Outcomes Study 36-Item Short Form Health Survey
Description: This survey is a generic health-related quality of life measure. Scores have normalized values with a mean of 50 and a standard deviation of 10, with higher scores indicating better health status. Results measure the average change in scores from baseline to follow-up.
Time Frame: Baseline, 3 months, and 12 Months post-surgery
Population: Women who completed the Medical Outcomes Study 36-Item Short Form Health Survey at baseline and 3 and 12 months after the index surgery.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Midurethral Sling | Sham Incision
Number analyzed (Participants) | 156 | 154
units on a scale
  3 Months - Mental Component | 1.5 (9.25) | 0.6 (8.44)
  3 Months - Physical Component | 2.1 (8.21) | 1.5 (7.52)
  12 Months - Mental Component: number analyzed (Participants) | 154 | 152
  12 Months - Mental Component | 1.9 (8.4) | 2.0 (8.94)
  12 Months - Physical Component: number analyzed (Participants) | 154 | 152
  12 Months - Physical Component | 3.1 (9.23) | 2.3 (7.51)

4. Secondary Outcome: Positive Cough Stress Test
Description: A leakage of urine with coughing or straining in either the supine or standing position with the bladder filled through a urethral catheter to 300 ml.
Time Frame: 3 and 12 Months Post-surgery
Population: Women who came in for 3 and 12 month post-op office visits and completed a cough stress test.
Measure: Count of Participants; unit: Participants
Arm/Group | Midurethral Sling | Sham Incision
Number analyzed (Participants) | 158 | 157
Participants
  3 Months | 10 | 54
  12 Months: number analyzed (Participants) | 143 | 151
  12 Months | 5 | 31

5. Secondary Outcome: Symptoms of Incontinence
Description: Symptoms that were at least moderately bothersome to the participant (as measured by a response of "moderately" or "quite a bit" to any of the four items on the Pelvic Floor Distress Inventory regarding leakage).
Time Frame: 3 and 12 Months Post-surgery
Population: Women who completed questions in the Pelvic Floor Distress Inventory regarding leakage 3 and 12 months after their index surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Midurethral Sling | Sham Incision
Number analyzed (Participants) | 160 | 165
Participants
  3 Months | 15 | 41
  12 Months: number analyzed (Participants) | 158 | 160
  12 Months | 18 | 30

6. Secondary Outcome: Treatment for Incontinence
Description: The need for treatment for any urinary incontinence, including surgery, medication, pessary for incontinence, supervised pelvic-muscle exercises, timed voiding and fluid management, periurethral injection, botulinum toxin injection, neuromodulation, or other treatment for incontinence.
Time Frame: 3 months post-surgery
Population: Women who reported whether or not they needed treatment for any urinary incontinence.
Measure: Count of Participants; unit: Participants
Arm/Group | Midurethral Sling | Sham Incision
Number analyzed (Participants) | 164 | 172
Participants | 11 | 13

7. Secondary Outcome: Pelvic Floor Distress Inventory (PFDI) Urinary Distress Inventory (UDI)
Description: PFDI is a symptom inventory for pelvic floor disorders. Scores ranges from 0 to 300, with higher scores indicating more symptoms. Results measure the average change in scores from baseline to follow-up.
Time Frame: Baseline, 3 months, and 12 months post-surgery
Population: Women who completed the PFDI UDI survey at baseline and 3 and 12 months after the index surgery.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Midurethral Sling | Sham Incision
Number analyzed (Participants) | 160 | 155
units on a scale
  3 Months | -44.9 (48.24) | -34.4 (44.92)
  12 Months: number analyzed (Participants) | 157 | 152
  12 Months | -43.1 (44.25) | -39.3 (40.93)

8. Secondary Outcome: Urinary Distress Inventory (UDI) Obstructive Symptom Subscale
Description: Scores on the UDI subscales range from 0 to 100, with higher score indicating more symptoms. Results measure the average change in scores from baseline to follow-up.
Time Frame: Baseline, 3 months, and 12 months post-surgery
Population: Women who completed the UDI obstructive symptom subscale survey at baseline and 3 and 12 months after the index surgery.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Midurethral Sling | Sham Incision
Number analyzed (Participants) | 160 | 158
units on a scale
  3 Months | -27.3 (22.69) | -28.0 (20.81)
  12 Months: number analyzed (Participants) | 157 | 154
  12 Months | -26.4 (22.69) | -27.1 (21.39)

9. Secondary Outcome: Urinary Distress Inventory (UDI) Irritative Symptom Subscale
Description: as for outcome 8
Time Frame: Baseline, 3 months, and 12 months post-surgery
Population: Women who completed the UDI irritative symptom subscale survey at baseline and 3 months after the index surgery.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Midurethral Sling | Sham Incision
Number analyzed (Participants) | 160 | 158
units on a scale
  3 Months | -12.5 (18.83) | -10.5 (17.06)
  12 Months: number analyzed (Participants) | 157 | 154
  12 Months | -10.9 (17.15) | -11.6 (15.87)

10. Secondary Outcome: Urinary Distress Inventory (UDI) Stress Subscale
Description: as for outcome 8
Time Frame: Baseline, 3 months, and 12 months post-surgery
Population: Women who completed the UDI stress subscale survey at baseline and 3 and 12 months after the index surgery.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Midurethral Sling | Sham Incision
Number analyzed (Participants) | 160 | 155
units on a scale
  3 Months | -5.1 (16.29) | 4.2 (20.42)
  12 Months: number analyzed (Participants) | 157 | 152
  12 Months | -5.7 (14.62) | -0.5 (16.89)

11. Secondary Outcome: Incontinence Severity Index
Description: Scores on the Incontinence Severity Index range from 1 to 12, with higher scores indicating greater severity. Results measure average change in scores from baseline.
Time Frame: Baseline, 3 months, and 12 months post-surgery
Population: Women who completed the Incontinence Severity Index survey at baseline and 3 and 12 months after the index surgery.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Midurethral Sling | Sham Incision
Number analyzed (Participants) | 157 | 156
units on a scale
  3 Months | -0.9 (3.01) | 0.6 (3.26)
  12 Months: number analyzed (Participants) | 154 | 152
  12 Months | -0.9 (2.7) | 0.1 (2.7)

ADVERSE EVENTS:
Time Frame: 12 months after index surgery
Arm/Group | Midurethral Sling | Sham Incision
Serious Adverse Events (participants affected / at risk) | 28/165 | 20/172
Other Adverse Events (participants affected / at risk) | 92/165 | 63/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Midurethral Sling (N=165) | Sham Incision (N=172)
Arrhythmia (Cardiac disorders) | 1 | 0
Congestive heart failure (Cardiac disorders) | 1 | 0
Pulse decreased (Investigations) | 1 | 0
Abnormal electrocardiogram (Investigations) | 1 | 0
Hypoxia (Injury, poisoning and procedural complications) | 0 | 1
Hypotension (Injury, poisoning and procedural complications) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Prolapse repair (Surgical and medical procedures) | 6 | 1
Appendicitis (Infections and infestations) | 2 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Rectocele repair (Surgical and medical procedures) | 1 | 0
Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Goitre (Endocrine disorders) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Mammogram abnormal (Investigations) | 0 | 1
Pain postoperative (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Pyelonephritis (Renal and urinary disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Vaginal haemorrhage postoperative (Injury, poisoning and procedural complications) | 1 | 2
Vaginal abscess (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Midurethral Sling (N=165) | Sham Incision (N=172)
Bladder perforation (Injury, poisoning and procedural complications) | 11/164 | 0
Urinary tract infection (Infections and infestations) | 49/158 | 30/164
Bladder retention at hospital discharge (Renal and urinary disorders) | 69/162 | 51/170
Bladder retention at 2 weeks (Renal and urinary disorders) | 9/163 | 1/169

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No